CLINICAL TRIAL: NCT05711979
Title: African American Resilient Caregivers
Acronym: AARC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COI disclosures
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00111805
Record Dates: First submitted 2023-01-19; First posted 2023-02-03 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2023-01

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AARC Intervention (Experimental): Participants in the AARC Intervention Arm will receive a 10 week intervention.
  Interventions: Behavioral: AARC

INTERVENTIONS:
Behavioral: AARC — There will be 10 90min weekly sessions. The first half of each session will consist of health education discussing diet, physical activity and screen time. Participants will set goals for themselves and their families. The investigators will check-in on goals and barriers to achieving goals in each session following the initial session. The second half of the sessions will focus on mindfulness based stress reduction including brief meditation, discussion of mindful eating and mindful parenting. This intervention will adapt an already-existing evidence-based obesity prevention program which has been administered to over 100 families (COACH), and it will add mindfulness-based stress reduction, tailored to African American women.

SUMMARY:
The purpose of this pilot study is to test the feasibility of a virtual intervention to prevent child obesity and cardiovascular disease in African American families.

DETAILED DESCRIPTION:
African American children experience a high prevalence of child obesity, increasing their subsequent risk of cardiovascular disease and diabetes. There is a lack of effective obesity prevention interventions for this population. Investigators also know that African American parents and caregivers experience high levels of stress and the manifestations of stress for African American women in particular may be unique and specific. Parent stress can lead to unhealthy family behaviors including less physical activity and a less healthy diet for parents and children. Given this background the investigators are creating a new intervention that combines an adapted evidence-based obesity prevention program (Competency Based Approach to Community Health - COACH) with mindfulness-based stress reduction tailored to African American women. As an initial step the investigators will pilot the intervention in a small number of African American women to determine whether the program is feasible.

ELIGIBILITY:
Inclusion Criteria:

* Identify as African American and female
* Have a child between the ages of 2-5 who lives with them at least 4 days per week that they care for as a parent or guardian.
* Feel comfortable discussing personal experiences and goals related to diet, PA, stress, parenting, etc. in front of a group of peers
* Access to zoom, preferably with video

Exclusion Criteria:

• Non English Speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 4 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Acceptability as assessed by semi-structured interviews | 10 weeks (post intervention)
  In this pilot study, acceptability of the intervention to the study population will be assessed by semi-structured interviews. Interview questions will identify features of the intervention which were beneficial to participants as well as barriers to participation.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle White, MD/MPH, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States